CLINICAL TRIAL: NCT02413957
Title: Pilot Project to Investigate the Influence of Medication Reconciliation and an Extensive Medication Safety Check on the Number of Adverse Drug Events in the Elderly
Brief Title: Medication Reconciliation in Comparison to an Extensive Medication Safety Check
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Ärztliche Zentrum für Qualität in der Medizin (Other); Universitätsklinikum Bonn - Institut für Patientensicherheit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14178
Record Dates: First submitted 2015-01-12; First posted 2015-04-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Elderly; Adverse Drug Event
Keywords: Elderly Patients; Medication Safety; Pharmaceutical Care; Medication Reconciliation
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Medication Reconciliation; Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Controll-Group (No Intervention): Patient randomized to the Control-Group will receive the traditional care by physician and nurse on the ward.
- MedRec-Group (Experimental): Patient randomized to the MedRec-Group will receive the traditional care by physician and nurse on the ward and additional pharmacist led medication reconciliation.
  Interventions: Other: Medication Reconciliation
- AMTS-Group (Experimental): Patient randomized to the AMTS-Group will receive the traditional care by physician and nurse on the ward and additional pharmaceutical care by a pharmacist.
  Interventions: Other: Pharmaceutical Care

INTERVENTIONS:
Other: Medication Reconciliation — Pharmacist take the best possible medication history (BPMH), comparison of the BPMH with the admission order (AMO), clarify and solve al discrepancies between the BPMH and the AMO.
  Arms: MedRec-Group
Other: Pharmaceutical Care — Checking medication under safety considerations (medication at admission, during hospital stay, at discharge); recommendations for inappropriate medication (e.g. contraindications or interactions) or medication related problems. Pharmaceutical care includes Medication Reconciliation.
  Arms: AMTS-Group

SUMMARY:
The purpose of this study is to determine wether an extensive medication safety check has a greater impact on the incidence of adverse drug events than medication reconciliation or no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient 65 years and older
* written informed consent patient or the legal representative
* existing medication therapy at hospitalization
* admission to one of the project wards via emergency department (non elective)

Exclusion Criteria:

- patients included in the study previously

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
incidence of adverse drug events | 1 year

SECONDARY OUTCOMES:
Assessment of the clinical relevance of medication related problems as determined by the French Society of Clinical Pharmacy | 1 year
  Severity scale for medication related problems: minor, significative, major, critical, catastrophic
Assessment of the clinical relevance of discrepancies as determined by the French Society of Clinical Pharmacy | 1 year
  Severity scale for discrepancies: minor, significative, major, critical, catastrophic
number of medication related problems | 1 year
number of discrepancies | 1 year
duration of taking the best possible medication history | 1 year
  The duration is measured in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aachen, Aachen, Germany

REFERENCES:
- [Background] Franzen K, Lenssen R, Jaehde U, Eisert A. [Medication Reconciliation-theory and practice]. Ther Umsch. 2014 Jun;71(6):335-42. doi: 10.1024/0040-5930/a000521. German. PMID 24867348